CLINICAL TRIAL: NCT07372768
Title: Lifting the Impacted Fetal Head; the Fetal Pillow and Tydeman Tube Trial
Acronym: LIFT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TCF 190908
Record Dates: First submitted 2025-12-11; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-12

CONDITIONS: Impacted Fetal Head; Full Dilatation Caesarean Section
Keywords: Impacted fetal head; Caesarean section; Full dilatation caesarean section; Tydeman Tube; Fetal Pillow

STUDY DESIGN:
Intervention Model Description: Sequential arms with 2 different treatments. 3-6 months using first device (Fetal Pillow), 3-6 months using second device (Tydeman Tube).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fetal Pillow (Active Comparator): The Fetal Pillow will be used for women undergoing full dilatation caesarean section who meet eligibillity criteria during the recruitment period of 3-6 months.
  Interventions: Device: Fetal Pillow
- Tydeman Tube (Active Comparator): The Tydeman tube will be used for women undergoing full dilatation caesarean section who meet eligibility criteria during the recruitment period of 3-6 months.
  In addition the Tydeman Tube will be used at the discretion of the operating clinician during caesarean sections performed at 7-9cm where an impacted fetal head is encountered unexpectedly.
  Interventions: Device: Tydeman Tube

INTERVENTIONS:
Device: Fetal Pillow — The Fetal Pillow is a CE marked single use sterile device. It is used in Caesarean sections performed at full dilatation. The Fetal Pillow is designed to atraumatically elevate the fetal head out of the pelvis before a caesarean section begins, making the delivery safer, easier and less traumatic. It comprises of a base plate, which is placed posteriorly in the vagina between the fetal head and the vaginal wall. It is then slowly inflated with 180mls of water via a thin tube, which aims to elevate the fetal head. It is removed at the end of the caesarean section.
  Some evidence for the Fetal Pillow suggests it can reduce maternal and fetal complications from FDCS by enabling elevation of a deeply engaged head, with some studies demonstrating a reduction in uterine incision extensions, lower estimated blood lossand fewer neonatal intensinve care (NICU)admissions. However evidence is conflicting and newer randomised control trials suggest no difference in outcome when using the device.
  Arms: Fetal Pillow
Device: Tydeman Tube — The Tydeman Tube is a UKCA/CE marked single use sterile device designed to aid delivery of an impacted fetal head at caesarean section. It consists of a semi-rigid wide bore silicone tube and flexible silicone cup.The tube is inserted into the vagina before or during caesarean section where an impacted fetal head is anticipated or encountered. It can be used from 7-10cm dilated. The cup fits against the baby's head. The tube is held by the assistant and used to elevate the head by pushing upwards. This disimpacts the head from the pelvis and brings it towards the surgeon's hand to enable delivery. The cup dissipates the force applied evenly over a wide area of the head which is intended to prevent fetal trauma. Once the surgeon has gained access below the head, the wide bore tube and design of the cup allows air to enter below the head during delivery to limit suction effect. Once the baby is delivered the Tydeman Tube is removed from the vagina.
  Arms: Tydeman Tube

SUMMARY:
A single centre prospective observational comparison trial to compare the Tydeman Tube and Fetal Pillow, to aid delivery of the impacted fetal head at full dilatation caesarean section, and to evaluate the use of the Tydeman Tube at 7-9cm.

DETAILED DESCRIPTION:
An impacted fetal head is a common complication encountered in 11% of all emergency caesarean sections and 65% of those performed at full dilatation. A recent UK Obstetric Surveillance Survey (UKOSS) highlighted significant maternal and neonatal complications secondary to an impacted fetal head, with 3% of babies dying or suffering a severe injury, and 6.1% of mother's requiring admission to intensive care, emphasizing the need to evaluate techniques and new devices to aid delivery. NHS resolution's early notification scheme implicated an impacted fetal head as a contributing factor in 9% of all severe neonatal brain injuries in 2019. There is no consensus amongst clinicians on the best management of an impacted fetal head, and with exponentially rising rates of intrapartum caesarean sections, improved management tools are urgently required.

This study will compare maternal and neonatal outcomes using two devices to aid delivery of an impacted fetal head at full dilatation caesarean section (FDCS)- the Tydeman Tube, a new UK Conformity Assessed (UKCA) and European Conformity (CE) marked device, and the Fetal Pillow, an existing CE marked device used commonly in clinical practice. There will be a separate observational sub study evaluating the use of the Tydeman Tube for managing an impacted fetal head at 7-9cm dilated. The study will also explore the acceptability of both devices to women and clinicians using postnatal questionnaires.

Participants will be all women requiring a full dilatation caesarean section who meet eligibility criteria. The study will be run in two consecutive arms - firstly, obstetricians and midwives will be trained to use the Fetal Pillow. The Fetal Pillow will then be introduced into clinical practice for 3-6 months. Following this the Fetal Pillow will be removed from clinical practice. Midwives and Obstetricians will then be trained to use the Tydeman Tube, which will be introduced into clinical practice for a further 3-6 months. During the Tydeman Tube arm of the trial, women undergoing caesarean section at 7-9cm who are found to have an impacted fetal head unexpectedly at the time of caesarean section are eligible for the observational sub study. If the operating surgeon believes the Tydeman Tube is required for the clinical situation then it may be used.

The trial is a prospective observational comparison trial with an additional observational sub study. The results of this study will be used to improve understanding on the best management techniques for an impacted fetal head.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing caesarean section at full dilataion for fetal pillow arm, or caesarean section at 7 or more centimetres dilated for the tydeman tube arm
* Singleton pregnancy
* Cephalic presentation

Exclusion Criteria:

* Allergy to silicone rubber
* Major congenital abnormalities
* Major anomaly of the fetal head (i.e. large encephalocele)
* Intrauterine death
* Suspected chorioamnionitis
* Active genital infection inc. Herpes Simplex Virus
* Cervical dilatation <10cm for fetal pillow arm and <7cm for tydeman tube arm
* Gestational age <37 weeks
* non-cephalic presentation

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Time from uterine incision to delivery | 4 weeks
  Seconds

SECONDARY OUTCOMES:
Uterine incision to closure time | 4 weeks
  Seconds
Estimated blood loss | 4 weeks
  mLs
Requirement of blood products | 4 weeks
  Yes/No
Volume of blood products | 4 weeks
  Dependent on type of product
Presence of uterine angle extensions | 4 weeks
  Yes/No
Presence of visceral injury | 4 weeks
  Yes/No - visceral injuries may include ureter, cervix, bladder, bowel
Need for hysterectomy | 4 weeks
  Yes/No
Presence of genital tract trauma | 4 weeks
  Yes/No - genital tract trauma may include lacerations and haematomas
Admission to HDU/ITU | 4 weeks
  Yes/No
Maternal death | 4 weeks
  Yes/No
Length of stay | 4 weeks
  Days
Wound infection | 4 weeks
  Yes/No
Endometritis | 4 weeks
  Yes/No
Change in maternal haemoglobin (Hb) | 4 weeks
  Difference in measured Hb before caesarean and after caesarean
Presence of birth trauma to the neonate | 4 weeks
  Yes/No - birth trauma may include intracranial haemorrhage, skull fracture, other fracture, facial nerve injury (bruising/facial nerve palsy/other nerve injury)
Apgar score | 4 weeks
  Routine test taken of the newborn infant based on Appearance (colour), Pulse (heart rate), Grimace (reflexes), Activity (muscle tone) and Respiration (breathing) at 5 and 10 minutes - scored from 0-10 with lower scores indicating poor condition and need for assessment/intervention
Resuscitation required | 4 weeks
  Yes/No
Admission to special care baby unit (SCBU) or neonatal intensive care unit (NICU) | 4 weeks
  Yes/No
Length of stay in higher care | 4 weeks
  Days
Arterial cord pH measurement | 4 weeks
  Measures the acidity of a newborn's blood from the umbilical artery, reflecting fetal oxygenation and metabolic state at birth, with normal ranges around 7.18-7.38, lower values (<7.0) can signal distress, risk of neurological issues and often require neonatal observation
Diagnosis of hypoxic-ischaemic encephalopathy (HIE) | 4 weeks
  Yes/No and Grading (1,2,3)
  HIE is a brain injury from lack of oxygen and/or blood flow to the brain around the time of birth, affecting newborns. It is associated with potential long-term disability including cerebral palsy or developmental delay, and in severe cases death. Symptoms include seizures, poor feeding and altered alternates. It is graded as mild (Grade 1), moderate (Grade 2) and severe (Grade 3)
Perinatal death | 4 weeks
  Yes/No
Neonatal feeding | 4 weeks
Evaluation of Fetal Pillow / Tydeman tube using Lickert scale questionnaires (clinician) | 4 weeks
  Acceptability, ease of use, perception of impacted head and perception of ease of delivery will be assessed using Lickert scale questionnaires where participants will be asked to rate their level of agreement or feeling on a symmetrical scale, form one extreme to another (i.e. 'strongly disagree' to 'strongly agree')
Acceptability of Fetal Pillow / Tydeman Tube using Lickert scan questionnaires (maternal) | 4 weeks
  Patients perception of the acceptability of the two devices will be assessed using Lickert scale questionnaires where participants will be asked to rate their level of agreement or feeling on a symmetrical scale, form one extreme to another (i.e. 'strongly disagree' to 'strongly agree')

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Shennan, MD, Principal Investigator — King's College London / Guy's and St Thomas'

IPD SHARING:
Plan to Share IPD: No